CLINICAL TRIAL: NCT03630315
Title: A Phase 1 Open-Label, Dose Escalation Study of OTX-TKI for Intravitreal Use in Subjects With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: CLN-0046: Treatment of AMD Subjects With OTX-TKI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0046
Record Dates: First submitted 2018-06-01; First posted 2018-08-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept; Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Low Dose) (Experimental): Subjects will receive a low dose of OTX-TKI
  Interventions: Drug: OTX-TKI
- Cohort 2 (Middle Dose) (Experimental): Subjects will receive a middle dose of OTX-TKI.
  Interventions: Drug: OTX-TKI
- Cohort 3 (High Dose) (Experimental): Subjects will receive a high dose of OTX-TKI.
  Interventions: Drug: OTX-TKI
- Cohort 3 (Anti-VEGF) (Experimental): Subjects will receive OTX-TKI plus a single anti-VEGF injection
  Interventions: Drug: OTX-TKI; Drug: Anti-VEGF
- Cohort 4 (High Dose) (Experimental): Subjects will receive a high dose of OTX-TKI.
  Interventions: Drug: OTX-TKI
- Cohort 4 (Anti-VEGF) (Experimental): Subjects will receive OTX-TKI plus a single anti-VEGF injection
  Interventions: Drug: OTX-TKI; Drug: Anti-VEGF

INTERVENTIONS:
Drug: OTX-TKI — OTX-TKI is a dried polyethylene glycol-based hydrogel fiber containing dispersed microcrystals of a small molecule tyrosine kinase inhibitor (TKI).
  Arms: Cohort 1 (Low Dose)
Drug: OTX-TKI — OTX-TKI is a dried polyethylene glycol-based hydrogel fiber containing dispersed microcrystals of a small molecule tyrosine kinase inhibitor (TKI).
  Arms: Cohort 2 (Middle Dose)
Drug: OTX-TKI — OTX-TKI is a dried polyethylene glycol-based hydrogel fiber containing dispersed microcrystals of a small molecule tyrosine kinase inhibitor (TKI).
  Arms: Cohort 3 (High Dose)
Drug: OTX-TKI — OTX-TKI is a dried polyethylene glycol-based hydrogel fiber containing dispersed microcrystals of a small molecule tyrosine kinase inhibitor (TKI).
  Arms: Cohort 3 (Anti-VEGF)
Drug: Anti-VEGF — Standard of care therapy used to block vascular endothelial growth factor
  Other Names: aflibercept; bevacizumab; ranibizumab
  Arms: Cohort 3 (Anti-VEGF)
Drug: OTX-TKI — OTX-TKI is a dried polyethylene glycol-based hydrogel fiber containing dispersed microcrystals of a small molecule tyrosine kinase inhibitor (TKI).
  Arms: Cohort 4 (Anti-VEGF); Cohort 4 (High Dose)
Drug: Anti-VEGF — Standard of care therapy used to block vascular endothelial growth factor
  Other Names: aflibercept; bevacizumab; ranibizumab
  Arms: Cohort 4 (Anti-VEGF)

SUMMARY:
To evaluate the safety, tolerability and efficacy of OTX-TKI for intravitreal use, in subjects who have neovascular age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
A multi-center, dose escalation, Phase 1, safety, tolerability and efficacy study to evaluate three dose groups of the OTX-TKI implant to treat subjects with a diagnosis of primary subfoveal neovascularization secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 50 years of age
* Are eligible for standard therapy
* Have active primary CNVM secondary to AMD, either newly diagnosed or previously treated with documented response to anti-VEGF therapy in the study eye [primary subfoveal CNV secondary to AMD including juxtafoveal lesions that affect the fovea] documented by FA and SD-OCT
* Are female who is postmenopausal for at least 12 months prior to screening or surgically sterile; or male or female of childbearing potential willing to use two forms of adequate contraception
* Are able and willing to comply with all study requirements and visits

Exclusion Criteria:

* Have previous laser photocoagulation to the center of the fovea in the study eye
* Have participated in any study involving an investigational drug either in the U.S. or outside the U.S. within the past 30 days
* Are an employee of the site that is directly involved in the management, administration, or support of the study, or be an immediate family member of the same
* Have a presence of a disease other than CNVM due to AMD in the study eye that could affect vision or safety assessments

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events for each subject | 9 months
  All adverse events from screening through end of study will be captured

SECONDARY OUTCOMES:
Determine the Maximum Tolerated Dose of the OTX-TKI injection | 9 months
  A Central Reading Center will evaluate multiple imaging modalities to confirm evidence of biological activity for subjects that have been treated with the OTX-TKI injection. If all subjects tolerate lower dosages, additional subjects will be treated at higher dosages. All data will be evaluated by the DSMC who, in concert with the Medical Monitor, will determine the Maximally Tolerated Dose.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Ocular Therapeutix, Inc., Sydney, Site 1
  - Ocular Therapeutiux, Inc., Sydney, Site 2
  - Ocular Therapeutiux, Inc., Sydney, Site 3
  - Ocular Therapeutix, Inc., Adelaide
  - Ocular Therapeutix, Inc., Albury
  - Ocular Therapeutix, Inc., Melbourne